CLINICAL TRIAL: NCT07314216
Title: A Single-Arm, Multicenter, Phase II Clinical Trial of Firmonertinib in Combination With Definitive Radiotherapy for Patients With Stage III Unresectable Pulmonary Adenocarcinoma Harboring Positive EGFR Uncommon Driver Mutations
Brief Title: Firmonertinib Combined With Definitive Radiotherapy in Stage III Unresectable EGFR Uncommon Mutant Pulmonary Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT172
Record Dates: First submitted 2025-11-25; First posted 2026-01-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: NSCLC (Non-small Cell Lung Carcinoma); Stage III; EGFR Uncommon Mutations
Keywords: unresectable Stage III lung adenocarcinoma; EGFR uncommon mutations; Firmonertinib; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Firmonertinib combined with definitive radiotherapy (Experimental): Patients in this arm will receive a combined regimen of Firmonertinib targeted therapy and definitive radiotherapy. The treatment consists of three phases:
  1. Induction Phase: Oral Firmonertinib monotherapy for 12 weeks;
  2. Combined Radiotherapy Phase: Firmonertinib concurrently with definitive thoracic radiotherapy for 6 weeks;
  3. Consolidation Phase: Firmonertinib monotherapy continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Firmonertinib; Radiation: Definitive Thoracic Radiotherapy

INTERVENTIONS:
Drug: Firmonertinib — Oral administration
  Other Names: AST2818
Radiation: Definitive Thoracic Radiotherapy — Conformal radiotherapy delivered to the primary tumor and involved regional lymph nodes.
  Other Names: IMRT; VMAT

SUMMARY:
This is a prospective, single-arm, Phase II clinical study aimed at evaluating the efficacy and safety of 160mg fimonertinib in combination with definitive radiotherapy for patients with EGFR uncommon driver mutation-positive, Stage III unresectable lung adenocarcinoma. The primary endpoint is Progression-Free Survival (PFS), assessed by the investigator according to RECIST 1.1 criteria, defined as the time from the first dose to objective disease progression or death (from any cause). Secondary endpoints include PFS by different mutation types, OS, ORR, DCR, as well as adverse events and their severity.

DETAILED DESCRIPTION:
The standard treatment for patients with unresectable Stage III non-small cell lung cancer (NSCLC) is definitive concurrent chemoradiotherapy followed by consolidative immunotherapy with durvalumab. However, the efficacy of this approach remains limited. For EGFR-mutant patients, the benefit of immunotherapy is modest, highlighting the need for alternative strategies. Although the third-generation EGFR-TKI firmonertinib has become a standard first-line therapy for advanced NSCLC harboring common EGFR mutations (exon 19 deletions and L858R), patients with uncommon EGFR mutations (e.g., G719X, S768I, L861Q, and various exon 20 insertion mutations) represent a heterogeneous and understudied population. For most of these uncommon mutations, no approved targeted therapy currently exists in the setting of Stage III unresectable NSCLC.

Firmonertinib is a novel, brain-penetrant third-generation EGFR-TKI that selectively and irreversibly inhibits both EGFR-sensitizing and T790M resistance mutations. It has demonstrated significant efficacy and a manageable safety profile in patients with EGFR T790M-mutant advanced NSCLC, and has also shown promising results in the first-line treatment of common EGFR mutations. Preclinical and clinical evidence suggests that combining EGFR-TKIs with radiotherapy may yield synergistic effects. Radiotherapy induces DNA damage and alters the tumor microenvironment, potentially enhancing both local and systemic efficacy of targeted agents. This combination strategy could be superior to sequential therapy or radiotherapy alone, particularly in molecularly selected populations. This study aims to explore the potential of this targeted-radiotherapy combination as a novel, chemotherapy-sparing, curative-intent treatment paradigm for patients with Stage III, EGFR uncommon mutation-positive lung adenocarcinoma.

This is an exploratory, Phase II, single-arm study. Enrolled patients will receive the study intervention consisting of oral firmonertinib (160 mg once daily) administered continuously until disease progression, unacceptable toxicity, or other treatment discontinuation criteria are met, concurrently with definitive radiotherapy. Radiotherapy will be delivered using intensity-modulated radiotherapy (IMRT) or volumetric modulated arc therapy (VMAT) to a total dose of 60 Gy in 30 fractions over approximately 6 weeks, with strict adherence to standard organ-at-risk dose constraints and institutional quality-assurance protocols. The primary objective is to evaluate progression-free survival (PFS). Secondary objectives include overall survival (OS), objective response rate (ORR), disease control rate (DCR), safety, and exploratory analyses within specific mutation subgroups.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study-specific procedures;
2. Age 18-75 years;
3. ECOG performance status of 0 or 1 with no deterioration within the 2 weeks prior to enrollment, and a life expectancy of ≥12 weeks;
4. Histologically or cytologically confirmed non-squamous non-small cell lung cancer;
5. Assessed as having unresectable or inoperable locally advanced non-squamous non-small cell lung cancer suitable for definitive radiotherapy (Stage III according to AJCC 9th edition TNM staging);
6. Presence of EGFR uncommon mutations (excluding 19del, L858R, T790M) confirmed by genetic testing in a tertiary grade A hospital; specific types are detailed in Appendix 11;
7. No prior systemic anti-tumor therapy or radiotherapy for locally advanced non-small cell lung cancer before the first dose of the study drug, including chemotherapy, biologic therapy, targeted therapy, immunotherapy, or investigational drug therapy;
8. At least one accurately measurable lesion according to RECIST 1.1, which has not been previously irradiated and was not biopsied during the screening period. If a subject has only one measurable lesion, biopsy of that lesion is permitted, provided the baseline imaging is performed at least 14 days after the biopsy;
9. Female subjects must use highly effective contraception (see restrictions) for at least 2 weeks prior to the first dose, have a negative pregnancy test, must not be breastfeeding at the time of treatment initiation, OR must meet at least one of the following criteria at screening to demonstrate the absence of childbearing potential;

   * Postmenopausal, defined as age over 50 years and amenorrhea for at least 12 months after cessation of all exogenous hormonal treatments;
   * For women aged 50 years or younger, amenorrhea for 12 months or more after cessation of exogenous hormone therapy and luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels within the institutional postmenopausal range;
   * Irreversible surgical sterilization documented by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but excluding tubal ligation;
10. Male subjects must be willing to use barrier contraception ;
11. Ability to comply with the study protocol and follow-up procedures, and capable of oral medication intake

Exclusion Criteria:

1. Pathological type is pulmonary squamous cell carcinoma or small cell lung cancer;
2. Known history of hypersensitivity to the active or inactive excipients of firmonertinib, or to drugs with a similar chemical structure or class to the investigational drug;
3. Confirmed presence of EGFR exon 19 deletion or exon 21 L858R mutation;
4. Presence of metastatic disease, or assessed as unsuitable for definitive radiotherapy; or unable to undergo definitive radiotherapy due to extensive tumor volume resulting in normal tissue radiation doses exceeding dose constraints;
5. NSCLC involving the superior sulcus, large cell neuroendocrine carcinoma (LCNEC), or sarcomatoid tumor;
6. Prior to the first dose of the study drug, patients who have received any of the following treatments;

   * Any prior EGFR-TKI therapy;
   * Patients who have received intrapleural infusion therapy; these patients may be enrolled only after pleural effusion has been stable for 28 days or more;
   * Major surgery within 28 days prior to the first dose of study drug (In China, major surgery is defined according to the Level 3 and Level 4 surgeries specified in the "Administrative Measures for the Clinical Application of Medical Technologies" implemented on May 1, 2009; see Appendix 5 for details);
   * Treatment with strong CYP3A4 inhibitors or inducers within 7 days prior to the first dose, or patients who require continued use of these drugs during the study period (see Appendix 6 for drug list);
   * Treatment with traditional Chinese medicine or Chinese patent medicine for anti-tumor indications within 7 days prior to the first dose, or patients who require continued use of these drugs during the study period;
   * Concurrent use of medications known to prolong the QTc interval or that may induce Torsade de Pointes, and which require continued administration during the study period (see Appendix 8 for drug list);
   * Discontinuation of other investigational drugs within less than 5 half-lives or 2 months (whichever is longer) prior to the first dose;
7. Toxicities from prior anti-tumor therapy have not recovered to ≤ CTCAE Grade 1 prior to the first dose of the study drug (except for alopecia or chemotherapy-induced peripheral neuropathy ≤ CTCAE Grade 2);
8. Patients with unstable pleural effusion;
9. History of, or diagnosis with, another malignancy within the past 5 years, except for effectively controlled basal cell carcinoma of the skin, carcinoma in situ of the cervix, and ductal carcinoma in situ of the breast;
10. Recent active digestive tract diseases, such as duodenal ulcer, ulcerative colitis, ileitis, etc.; intestinal perforation; intestinal fistula; or other conditions deemed by the investigator as potentially leading to gastrointestinal bleeding or perforation; or refractory nausea/vomiting, chronic gastrointestinal diseases, inability to swallow the study drug, or prior extensive bowel resection that would preclude adequate absorption of firmonertinib;
11. Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension, diabetes, active bleeding, etc., which in the investigator's judgment is not conducive to the patient's participation in the study or may compromise protocol compliance; or active infection including Hepatitis B, Hepatitis C, and Human Immunodeficiency Virus (HIV) (including any patient receiving intravenous treatment for infection; active hepatitis B infection at a minimum includes all patients serologically positive for HBsAg with HBV DNA >1000 copies/mL);
12. History of interstitial lung disease (ILD), drug-induced ILD, prior history of radiation pneumonitis requiring steroid treatment, or any evidence of active ILD;
13. Any known evidence of corneal lesions/damage;
14. Inadequate bone marrow reserve or organ function based on examinations within 28 days prior to the first dose of study drug (without transfusion or blood products, granulocyte colony-stimulating factor, or other hematopoietic stimulators within 2 weeks prior to testing);

    * Absolute neutrophil count <1.5 × 10^9/L; Platelet count <100 × 10^9/L; Hemoglobin <90 g/L;
    * Alanine aminotransferase > 2.5 × ULN; Aspartate aminotransferase >2.5 × ULN; Total bilirubin > 1.5 × ULN, or for patients with liver metastases, AST and/or ALT >5 × ULN;
    * Serum creatinine >1.5 × ULN, OR Creatinine clearance <50 mL/min (measured or calculated using the Cockcroft and Gault formula, see Appendix 2);
    * International Normalized Ratio > 1.5, AND Activated Partial Thromboplastin Time >1.5 × ULN;
15. Any of the following cardiac criteria;

    * Mean resting corrected QT interval (QTc) >470 msec obtained from 3 consecutive ECGs, calculated using Fridericia's formula;
    * Any clinically significant abnormalities in rhythm, conduction, or morphology of resting ECG within 28 days prior to the first dose, e.g., complete left bundle branch block, third-degree, and second-degree heart block;
    * Cardiac function assessment within 28 days prior to the first dose: Left Ventricular Ejection Fraction <50%; history of myocardial infarction, severe/unstable angina, or coronary artery bypass graft surgery within the past 6 months; or cardiac insufficiency ≥ NYHA Class 2;
16. Pregnancy or lactation;
17. Patients judged by the investigator as ineligible for the study, such as those unlikely to comply with the study protocol, procedures, and requirements; or any other circumstances warranting exclusion based on the investigator's discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From enrollment until 30 months after the completion of treatment
  the time from the first dose of study treatment (or treatment initiation in single-arm trials) to disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate | From enrollment until 30 months after the completion of treatment
  Investigator-assessed objective response rate (complete response + partial response) per RECIST v1.1
Disease control rate | From enrollment until 30 months after the completion of treatment
  Investigator-assessed objective response rate (complete response + partial response) per RECIST v1.1
Progression-Free Survival by Mutation Type | From enrollment until 30 months after the completion of treatment
  Investigator-assessed (per RECIST v1.1) time from first study treatment to objective disease progression or death from any cause, by mutation type
Overall Survival | From enrollment until 60 months after the completion of treatment
  Investigator-assessed time from the first dose of study treatment to death from any cause
AE | From enrollment until 30 months after the completion of treatment, every 12 weeks
  Investigator-assessed by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Huai Liu, M.Med., Principal Investigator — Hunan Cancer Hospital; Xingxiang Pu, M.D., Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No